CLINICAL TRIAL: NCT05777746
Title: The Effect of an Online Plant-Based Dietary Program on Cardiovascular Risk Factors in Persons With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Acronym: Plate-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, dr.Frank L.J. Visseren, professor doctor F.L.J. Visseren, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL80378.041.22
Record Dates: First submitted 2022-12-27; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Diet, Vegetarian; Diet, Vegan; Cardiometabolic Risk Factors; Cholesterol, LDL; Blood Pressure; Glycemic Control; Diet Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: An investigator and outcome assessor blinded design is chosen to reduce bias. All investigators collecting data by physical examination will be blinded to the allocation of the patients. Similarly, lab technicians performing the blood measurements will be blinded to the patient allocation. Lastly, the statistical analyses will be performed blinded to the allocation of patient groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An online 12 week plant-based dietary program (Experimental)
  Interventions: Behavioral: 12-week plant-based dietary program
- Usual Diet (Other)
  Interventions: Behavioral: Usual Diet

INTERVENTIONS:
Behavioral: 12-week plant-based dietary program — a 12-week plant-based dietary program consisting of information via an online platform, online guidance by dieticians and in online peer support groups. Patients will aim to maximize their intake of plant-based products while reducing their of animal products as much as possible.
  Arms: An online 12 week plant-based dietary program
Behavioral: Usual Diet — Patients in the control group continue with their usual diet and/or usual dietary care. Patients in the control group will be offered access to the online platform at 24 weeks.
  Arms: Usual Diet

SUMMARY:
Persons with Type 2 Diabetes (T2D) are at an increased risk of cardiovascular disease (CVD) and mortality. Dietary changes are recommended by guidelines to treat T2D and reduce risk of CVD. Plant-based diets eliminate certain (i.e. vegetarian diet) or eliminate all animal based products (i.e. vegan diet). Clinical trials with plant-based diets have not looked at incidence of CVD as a (primary) outcome, but at intermediate outcomes of cardiovascular risk. A meta-analysis of 8 trials including 369 persons with T2D found an effect of a plant-based diet on glycated hemoglobin (HbA1c) of -0.29% [95% CI: -0.45, -0.12%] relative to mostly (omnivorous) low-fat diets or usual diet. The 95%CI ranged from what the authors had defined as clinically trivial to clinically relevant. For lipids, a network meta-analysis in persons with T2D compared the effect of a plant-based diet to a (omnivorous) low fat diet (274 patients allocated to a plant-based diet vs 2047 patients allocated to low fat diets). Compared to omnivorous low fat diets, the mean effect of plant-based diets on LDL-Cholesterol was -0.33 mmol/L [95%CI:- 0.55, - 0.12]. However, the quality of the evidence for this estimate was graded as low, mainly due to imprecision and within-study-bias. Furthermore, plant-based diets might reduce blood pressure (BP). However, while vegetarian diets reduce BP in patients with and without hypertension, for vegan diets the effect was only significant in patients with a systolic BP>130mmHgz (see section 1.4.3). Additionally, the effect of plant-based diets on inflammation, which might also be causally related to CVD risk in persons with T2D, has not been reported in trials with persons with T2D. Furthermore, most clinical trials of plant-based diets in persons with T2D have used resource intensive interventions, like weekly group meetings and cooking sessions. The effect of an online plant-based dietary intervention, which is more scalable, has not been reported in clinical trials. Lastly, factors influencing adherence in these trials have not been reported.

In summary, plant-based diets likely lower CVD risk by lowering HbA1c, LDL cholesterol and potentially blood pressure in persons with T2D. However, estimated effect sizes are imprecise and the effect on inflammation is still unknown. Furthermore, trials to date have used resource intensive interventions. Thus, the present trial aims to study the effect of a primarily online plant-based dietary program on (cardio)vascular risk factors in persons with T2D. Additionally, adherence and factors influencing adherence will be investigated. Participants will be randomized to the intervention or control group. The intervention group will be guided to transition to a plant-based dietary pattern using an online platform and online sessions. Researchers will compare the intervention group to the control group, that continues with usual diet, to see if the cardiovascular risk profile of the intervention group improves.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of Type 2 Diabetes made by a physician
2. Using oral glucose-lowering medication and/or an insulin regime with a stable dose during at least the last two months before the screening visit;
3. Diagnosis of type 2 diabetes was made more than one year ago
4. Age of 18 years or older on the day of signing the informed consent form.
5. When the patients is also using lipid-lowering and/or blood pressure-lowering medication, than the dose should be stable for at least two months before the screening.

Exclusion criteria

1. Insulin-dependent type 2 diabetes in combination with hypoglycemia unawareness. Hypoglycemia unawareness is defined as the onset of hypoglycemia before the appearance of autonomic symptoms or failure to recognize hypoglycemia.
2. Two or more episodes of severe hypoglycemia (glucose < 3 mmol/L) during the last 3 months;
3. Uncontrolled T2D, defined as a HbA1c >86 mmol/mol (>10%);
4. Uncontrolled hypertension, defined as an office systolic blood pressure ≥ 180mmHg;
5. Inability to attend at least 60% of the scheduled meetings;
6. Pregnancy or a wish to get pregnant during the study period;
7. Diagnosis of familial hypercholesterolemia;
8. Being diagnosed with osteoporosis.
9. Known vitamin B12 deficiency, defined as serum vitamin B12 <130 pmol/L or using vitamin B12 supplements prescribed by a physician;
10. Known iron deficiency defined as a serum ferritin < 25µg/L for males or < 20µg/L for females or using iron supplements prescribed by a physician;;
11. The presence of any disease for which the patients uses a specific diet and where transitioning to a plant-based diet might lead to unfavorable effects on this disease as judged by the research team and/or the treating physician. An exception is a salt-restricted diet for hypertension;
12. Current or planned participation in any other interventional study within 30 days of signing the informed consent form;
13. Any medical, social or physiological circumstance which might interfere with the study, based on judgement by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c (mmol/mol) | Week 12
Composite of Estimated relative CVD risk (based on change in LDL-c , SBP and HbA1c) | Week 12

SECONDARY OUTCOMES:
Calculated absolute CVD risk reduction (%) | Week 12, 24 and 36
  Using baseline parameters (e.g. baseline LDL-C, BP, HbA1c, manifest CVD, duration of diabetes) and the risk prediction model DIAL2/SCORE-2(OP), the absolute CVD risk at baseline is calculated. The expected absolute risk reduction is calculated using changes in CVD risk profile after 12 and 24 weeks
HbA1c and estimated change in absolute and relative CVD risk (based on change in LDL-c, SBP and HbA1c) | Week 12, 24 and 36
  Per-protocol analysis
Glycemic control (HOMA2-IR, HOMA2-B%, TyG-index, NAFLD Score) | Week 12 and 24
Lipids and lipoprotein profile | Week 12 and 24
  Composition and concentration of lipoproteins and lipids, including total cholesterol, HDL-cholesterol, apolipoprotein-B, LDL-C and triglycerides
Blood pressure (systolic and diastolic) | Week 12 and 24
Inflammatory profile (CRP, neutrophil and lymphocyte count) | Week 12 and 24
Quality of life(EQ-5D, self-perceived stress,and DDRQOL-R(-9), medication use) | Week 12 and 24
Anthropometric measurements (BMI, hip/waist ratio) | Week 12, 24 and 36
Adherence (dietary index) | Week 12, 24 and 36
Rate of Vitamin B12 and ferritin deficiency | Week 12 and 24

OTHER OUTCOMES:
Subgroup analysis | Week 12 and 24
  Subgroups will be made on the basis of baseline characteristics (e.g. age, level of education, gender, presence of hypertension, duration of T2D, use of insulin, BMI, HbA1c)
Effect modification by diabetes subtype and adherence to the plant-based diet | Week 12 and 24
Determinants of adherence | Week 12 and 24
  Patient characteristics
Determinants of adherence | Week 12 and 24
  Based on outcome of the Food Choice questionnaire
Determinants of adherence | Week 12 and 24
  Based on outcome of the Self-Efficacy questionnaire
Determinants of adherence | Week 12 and 24
  Based on outcome of the in-group identification questionnaire
Effect of the 12-week online dietary program on the CVD risk profile in the control group | Week 36
Incident Hypoglycemia | Week 12 and 24
  Incidence of mild and severe hypoglycemia
Physical Activity (Metabolic Equivalent Tasks) | Week 12 and 24
  Measured using the SQUASH questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Medicine UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Request for IPD should be directed to the PI. The PI will judge whether request are appropriate and can be granted within the existing rules and regulations.

REFERENCES:
- See also: Plate-DM UMC Utrecht — https://www.umcutrecht.nl/nl/wetenschappelijk-onderzoek/plate-dm